CLINICAL TRIAL: NCT01538511
Title: A Two-centre, Randomised, Open-labelled, Four-week, Parallel-group Pharmacokinetics Trial in Japanese Type 2 Diabetic Subjects Characterising the Insulin Profile of Thrice Daily Regimen With Biphasic Insulin Aspart 70 (NN2000-Mix70) With Reference to That of Twice Daily Regimen With Biphasic Insulin Aspart 30 (NN-X14Mix30) and Physiological Insulin Profile in Japanese Healthy Volunteers
Brief Title: Insulin Profile of Biphasic Insulin Aspart 70 to That of Biphasic Insulin Aspart 30 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1638
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 70 (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 70 — Administered subcutaneously (s.c., under the skin) three times daily immediately before breakfast, lunch and dinner for 4 weeks. Dose individually adjusted
  Arms: BIAsp 70
Drug: biphasic insulin aspart 30 — Administered subcutaneously (s.c., under the skin) twice daily immediately before breakfast and dinner for 4 weeks. Dose individually adjusted
  Arms: BIAsp 30

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to compare biphasic insulin aspart 70 (NN2000-Mix70) in subjects with type 2 diabetes with that of biphasic insulin aspart 30 (NN-X14Mix30) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

SUBJECTS WITH TYPE 2 DIABETES

* Subjects with type 2 diabetes mellitus
* Current treatment using intermediate-acting, long-acting or pre-mixed/biphasic insulin preparation (including insulin analogues) in once or twice daily (before breakfast and dinner) treatment regimen for at least 12 weeks (a temporary use [maximum of one week in total] of rapid-acting human insulin will be allowed)
* Age between 20-69 years, both inclusive
* HbA1c (glycosylated haemoglobin A1c) below 9.0%
* Body Mass Index (BMI) 18.5-25.0 kg/m^2
* Total daily insulin dose (per day) above 0.2 U or IU/kg body weight and below 1.0 U or IU/kg body weight HEALTHY VOLUNTEERS
* Japanese subjects with considered generally healthy based on medical history and physical examination
* Age between 20-29 years, both inclusive
* Body Mass Index (BMI) 18.5-25.0 kg/m^2
* Subjects with normal glucose tolerance (NGT); defined as fasting plasma glucose below 110 mg/dL and 2-hour post OGTT (oral glucose tolerance test) plasma glucose below 140 mg/dL

Exclusion Criteria:

SUBJECTS WITH TYPE 2 DIABETES

* Proliferative retinopathy or maculopathy requiring acute treatment
* Impaired hepatic function
* Impaired renal function
* Serious cardiac diseases
* Uncontrolled hypertension
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia
* Current treatment or expected at the screening to start treatment with systemic corticosteroids HEALTHY VOLUNTEERS
* Any clinical laboratory values deviated from the reference range at the laboratory (except for cases within physiological change) at the screening
* History or presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* Subjects with a first-degree relative with diabetes mellitus

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-06-05 (Actual); Primary Completion 2007-03-13 (Actual); Study Completion 2007-03-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma insulin concentration curve from 0 to 24 hours

SECONDARY OUTCOMES:
Area under the concentration curve of plasma insulin from 0 to 4 hours after meals
Maximum plasma insulin concentration observed from 0 to 4 hours after meals
Time to reach the maximum plasma insulin concentration from 0 to 4 hours after meals
The 24-hour plasma insulin profile deviances in Japanese type 2 diabetic subjects
Pre-meal plasma glucose concentration before meals
Postprandial plasma glucose (PPPG) excursion from 0 to 4 hours after meals
The maximum plasma glucose concentration observed from 0 to 4 hours after meals
The time to reach the maximum plasma glucose concentration of observed from 0 to 4 hours after meals
Average of plasma glucose concentration from 0 to 24 hours
The area under the plasma C-peptide concentration curve from 0 to 24 hours derived from the 24-hour plasma C-peptide profile
Frequency of hypoglycaemic episodes
Frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com